CLINICAL TRIAL: NCT05361278
Title: Evaluation of Irrigation Effectiveness for Gel and Solution of Chlorhexidine in Disinfection Root Canals of Primary Anterior Teeth.
Brief Title: Evaluation of Gel and Solution of Chlorhexidine in Disinfection Root Canals of Primary Anterior Teeth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-Pedo-02-2022
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Dental Caries; Infection, Bacterial; Tooth, Deciduous
Keywords: Anterior Primary Tetth; Infected canals; chlorhexidine; Sodium hypochlorite
MeSH Terms: conditions — Dental Caries; Bacterial Infections | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chlorhexidine irrigation solution (Experimental): CHx 2% solution will be used.
  Interventions: Other: Chlorhexidine solution
- Activated chlorhexidine irrigation solution (Experimental): CHx 2% solution will be used with ultrasonic activation.
  Interventions: Other: Activated chlorhexidine solution
- Chlorhexidine irrigation gel (Experimental): CHx 2% gel will be used.
  Interventions: Other: Chlorhexidine gel
- Activated chlorhexidine irrigation gel (Experimental): CHx 2% gel will be used with ultrasonic activation.
  Interventions: Other: Activated chlorhexidine gel
- Sodium hypochlorite irrigation solution (Other): NaOCl 5,25% solution will be used.
  Interventions: Other: Sodium hypochlorite solution

INTERVENTIONS:
Other: Chlorhexidine solution — * Irrigate the root canal with 1 ml of 2% CHx solution between each file 1 mm from the apical foramen by using a 27-gauge irrigation needle.
  * Irrigate the root canal with 3 ml of the solution after using the last file.
  * Irrigation with 3 ml of 0.5% Tween 80 and 0.07 % lecithin to remove residual chlorhexidine solution.
  * Drying the canal with paper points (placing a 20 size paper point for 60 seconds in each canal) to take the bacterial smear.
  * Follow-up of endodontic treatment procedures for the treated tooth.
  Arms: Chlorhexidine irrigation solution
Other: Activated chlorhexidine solution — * Irrigate the root canal with 1 ml of 2% CHx solution between each file 1 mm from the apical foramen by using a 27-gauge irrigation needle with activation using an ultrasonic irrigation head.
  * Irrigate the root canal with 3 ml of the solution after using the last file with activation using an ultrasonic irrigation head.
  * Irrigation with 3 ml of 0.5% Tween 80 and 0.07 % lecithin to remove residual chlorhexidine solution.
  * Drying the canal with paper points (placing a 20 size paper point for 60 seconds in each canal) to take the bacterial smear.
  * Follow-up of endodontic treatment procedures for the treated tooth.
  Arms: Activated chlorhexidine irrigation solution
Other: Chlorhexidine gel — * Irrigate the root canal with 1 ml of 2% CHx gel between each file 1 mm from the apical foramen by using a 27-gauge irrigation needle.
  * Irrigate the root canal with 3 ml of the gel after using the last file.
  * Irrigation with 3 ml of 0.5% Tween 80 and 0.07 % lecithin to remove residual chlorhexidine gel.
  * Drying the canal with paper points (placing a 20 size paper point for 60 seconds in each canal) to take the bacterial smear.
  * Follow-up of endodontic treatment procedures for the treated tooth.
  Arms: Chlorhexidine irrigation gel
Other: Activated chlorhexidine gel — * Irrigate the root canal with 1 ml of 2% CHx gel between each file 1 mm from the apical foramen by using a 27-gauge irrigation needle with activation using an ultrasonic irrigation head.
  * Irrigate the root canal with 3 ml of the gel after using the last file with activation using an ultrasonic irrigation head.
  * Irrigation with 3 ml of 0.5% Tween 80 and 0.07 % lecithin to remove residual chlorhexidine gel.
  * Drying the canal with paper points (placing a 20 size paper point for 60 seconds in each canal) to take the bacterial smear.
  * Follow-up of endodontic treatment procedures for the treated tooth.
  Arms: Activated chlorhexidine irrigation gel
Other: Sodium hypochlorite solution — * Irrigate the root canal with 1 ml of 5.25% sodium hypochlorite solution between each file 1 mm from the apical foramen by using a 27-gauge irrigation needle.
  * Irrigate the root canal with 3 ml of the solution after using the last file.
  * Irrigating the canal with 3 ml of 5% sodium thiosulfate solution to remove residual of sodium hypochlorite.
  * Drying the canal with paper points (placing a 20 size paper point for 60 seconds in each canal) to take the bacterial smear.
  * Follow-up of endodontic treatment procedures for the treated tooth.
  Arms: Sodium hypochlorite irrigation solution

SUMMARY:
The process of removing bacteria and their products from the root canals is an essential step that is achieved through the combination of mechanical preparation and irrigation with chemicals. However, mechanical preparation alone can not reduce the microbial formations inside root canals, so at least about 35% of the root canal walls remain without the preparation tools reaching them.

Many irrigants were used to irrigate the root canals, as sodium hypochlorite and chlorhexidine are the most famous. Although most studies have proven the effectiveness of sodium hypochlorite with its different concentrations in accomplishing this task, some of them showed the inability of the irrigant fluid to eliminate Enterococcus faecalis inside the canals. These bacteria are highly resistant, and therefore endodontic treatment fails in the long term.

DETAILED DESCRIPTION:
Bacteria and their products play an essential role in the initiation and persistence of endodontic diseases. Therefore, eliminating them and preventing the return of their effectiveness is the desired goal in any successful endodontic treatment in the short and long term.

Due to the fact that mechanical preparation of the root canal alone is not capable of removing the entire bacterial content, chemical irrigants were considered necessary to reduce the number of bacteria and toxins resulting from them. Until now, there is no irrigant capable of removing the entire bacterial content from the root canal.

Despite the many advantages of sodium hypochlorite, several studies have revealed the toxicity of the solution in high concentrations of it, and it tends to cause tissue irritation when it comes into contact with the apical tissues.

Chlorhexidine has been used for a long time in dentistry due to its antibacterial properties, long period of effect, and relatively low toxicity. This has prompted its use as an irrigant and an intra-canal dressing in endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Definitely positive or positive ratings of Frank scale.
2. Physiological root resorption no more than the apical third
3. Symptoms or signs of pulpal necrosis with or without radial lesions (swelling - fistua - abnormal movement).
4. At least 2 mm of bone surrounding the permanent bud.
5. Children who have not taken antibiotics in the past 3 months.

Exclusion Criteria:

1. Systematic or mental disorders.
2. Definitely negative or negative ratings of Frankel scale
3. Existence external or internal abnormal absorption.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Logarithmic reduction of bacterial count within the root canal of chlorhexidine solution. | 24 hours after sample incubation
  Set the Petri dish on a grid background and count the colonies in each grid cell, moving in a methodical pattern through all of the cells.
Logarithmic reduction of bacterial count within the root canal of activated chlorhexidine solution. | 24 hours after sample incubation
  Set the Petri dish on a grid background and count the colonies in each grid cell, moving in a methodical pattern through all of the cells.
Logarithmic reduction of bacterial count within the root canal of chlorhexidine gel. | 24 hours after sample incubation
  Set the Petri dish on a grid background and count the colonies in each grid cell, moving in a methodical pattern through all of the cells.
Logarithmic reduction of bacterial count within the root canal of activated chlorhexidine gel. | 24 hours after sample incubation
  Set the Petri dish on a grid background and count the colonies in each grid cell, moving in a methodical pattern through all of the cells.
Logarithmic reduction of bacterial count within the root canal of sodium hypochlorite solution. | 24 hours after sample incubation
  Set the Petri dish on a grid background and count the colonies in each grid cell, moving in a methodical pattern through all of the cells.

CONTACTS AND LOCATIONS:
Overall Officials: Rahaf ِA kharsa, DDs, Principal Investigator — MSc student in Pedodontics, University of Damascus; Mohannad G Laflouf, Phd, Study Director — Professor of Pedodontics, Department of Pedodontics, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goud S, Aravelli S, Dronamraju S, Cherukuri G, Morishetty P. Comparative Evaluation of the Antibacterial Efficacy of Aloe Vera, 3% Sodium Hypochlorite, and 2% Chlorhexidine Gluconate Against Enterococcus faecalis: An In Vitro Study. Cureus. 2018 Oct 22;10(10):e3480. doi: 10.7759/cureus.3480. PMID 30648031
- [Background] Gomes BP, Ferraz CC, Vianna ME, Berber VB, Teixeira FB, Souza-Filho FJ. In vitro antimicrobial activity of several concentrations of sodium hypochlorite and chlorhexidine gluconate in the elimination of Enterococcus faecalis. Int Endod J. 2001 Sep;34(6):424-8. doi: 10.1046/j.1365-2591.2001.00410.x. PMID 11556507
- [Background] Ruksakiet K, Hanak L, Farkas N, Hegyi P, Sadaeng W, Czumbel LM, Sang-Ngoen T, Garami A, Miko A, Varga G, Lohinai Z. Antimicrobial Efficacy of Chlorhexidine and Sodium Hypochlorite in Root Canal Disinfection: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Endod. 2020 Aug;46(8):1032-1041.e7. doi: 10.1016/j.joen.2020.05.002. Epub 2020 May 12. PMID 32413440
- [Background] Walia V, Goswami M, Mishra S, Walia N, Sahay D. Comparative Evaluation of the Efficacy of Chlorhexidine, Sodium Hypochlorite, the Diode Laser and Saline in Reducing the Microbial Count in Primary Teeth Root Canals - An In Vivo Study. J Lasers Med Sci. 2019 Fall;10(4):268-274. doi: 10.15171/jlms.2019.44. Epub 2019 Oct 1. PMID 31875118
- [Background] Tirali RE, Bodur H, Ece G. In vitro antimicrobial activity of sodium hypochlorite, chlorhexidine gluconate and octenidine dihydrochloride in elimination of microorganisms within dentinal tubules of primary and permanent teeth. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e517-22. doi: 10.4317/medoral.17566. PMID 22143724